CLINICAL TRIAL: NCT02431650
Title: A Proof-Of-Concept Study to Assess the Effectiveness of OZ439 as a Gametocytocidal and Transmission Blocking Agent in Experimental P. Falciparum Infection
Brief Title: Effectiveness of OZ439 as a Gametocytocidal and Transmission Blocking Agent
Acronym: OZGAM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Q-Pharm Pty Limited (Industry); Clinical Network Services (CNS) Pty Ltd (Industry); Sullivan Nicolaides Pathology (Industry); QIMR Berghofer Medical Research Institute (Other); Army Malaria Institute, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QP15C05
Record Dates: First submitted 2015-04-17; First posted 2015-05-01 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Malaria
Keywords: Induced blood stage malaria; Transmission; Mosquito feeding; OZ439; Primaquine; Piperaquine; Artefonomel
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OZ439 (Experimental): Each participant in the cohort will be inoculated on Day 0 with ~2,800 viable parasites of Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. when PCR quantification of all participants is ≥ 5,000 parasites/mL, they will receive a single dose of 480 mg of piperaquine phosphate to clear blood stage parasitemia. When gametocytemia is at the peak (approximately 15 days after administration of piperaquine), participants will be randomised to receive either OZ439 or a control group (primaquine treatment).
  In the first cohort 500 mg OZ439 will be administered as a single dose. Doses used in subsequent cohort(s) will be determined following a review of observed safety and pharmacodynamic drug effects.
  Interventions: Drug: OZ439
- Primaquine (Active Comparator): Each participant in the cohort will be inoculated on Day 0 with ~2,800 viable parasites of Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. when PCR quantification of all participants is ≥ 5,000 parasites/mL, they will receive a single dose of 480 mg of piperaquine phosphate to clear blood stage parasitemia. When gametocytemia is at the peak (approximately 15 days after administration of piperaquine), participants will be randomised to receive either OZ439 or a control group (primaquine treatment).
  Primaquine is a positive control for OZ439, to be administered 15 mg as a single dose.
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: OZ439
  Other Names: Artefonomel
  Arms: OZ439
Drug: Primaquine
  Arms: Primaquine

SUMMARY:
This is a single-centre, controlled, open label study using P. falciparum-induced blood stage malaria (IBSM) infection to assess the effectiveness of OZ439 as a gametocytocidal agent, as well as its treatment effects on gametocyte infectivity and development in vector mosquitoes. Previous clinical studies including one IBSM study have shown that in addition to effectively clearing replicating, asexual (pathogenic) life cycle stages of malaria, a single dose of piperaquine (480 mg) results in the production of gametocytes, as determined by gametocyte-specific transcript (pfs25) qPCR. The propensity of piperaquine to induce gametocytaemia will be employed in this study to assess the efficacy of OZ439 as a gametocytocidal and transmission blocking agent. Experimental mosquito feeding via both direct feeding on participants and artificial (indirect) membrane mosquito feeding will be performed. The study will be conducted in up to 3 cohorts where participants will be randomised into an experimental or a control group (n=2 per group) when peak gametocytemia occurs (approximately 15 days after administration of piperaquine).

DETAILED DESCRIPTION:
This is a single-centre, controlled, open label study using P. falciparum-induced blood stage malaria (IBSM) infection to assess the effectiveness of OZ439 as a gametocytocidal agent, as well as its treatment effects on gametocyte infectivity and development in vector mosquitoes. Previous clinical studies including one IBSM study have shown that in addition to effectively clearing replicating, asexual (pathogenic) life cycle stages of malaria, a single dose of piperaquine (480 mg) results in the production of gametocytes, as determined by gametocyte-specific transcript (pfs25) qPCR. The propensity of piperaquine to induce gametocytaemia will be employed in this study to assess the efficacy of OZ439 as a gametocytocidal and transmission blocking agent. Experimental mosquito feeding via both direct feeding on participants and artificial (indirect) membrane mosquito feeding will be performed. The study will be conducted in up to 3 cohorts where participants will be randomised into an experimental or a control group (n=2 per group) when peak gametocytemia occurs (approximately 15 days after administration of piperaquine). The groups will be of equal size with participants in the experimental group receiving OZ439 and participants in the control group receiving primaquine (positive control for OZ439, to be administered 15 mg as a single dose). The dose of OZ439 that will be investigated in the experimental group of the first cohort will be 500 mg administered as a single dose. Doses used in subsequent cohort(s) will be determined following a review of observed OZ439 safety, and pharmacodynamic drug effects as defined by gametocyte clearance kinetics and transmission blocking activity. The doses used in cohort 2 and 3 may be adjusted, but will not exceed the maximum acceptable dose predefined for this study (i.e. 1200 mg OZ439) as determined in previous safety and pilot efficacy studies. The dose will be determined by the funding sponsor and the principal investigator (PI) following Safety Review team (SRT) and scientific evaluation. Subsequent cohorts will not commence until at least after day 28 of the previous cohort and review by Safety Review Team. This interval will also allow cohorting of experimental infection of mosquitoes to optimise logistics and enable iterative improvements in the system if applicable.

Each participant in the cohort will be inoculated on Day 0 with ~2,800 viable parasites of Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. On an outpatient basis, participants will be monitored daily via phone call and then daily (AM) from day 4 (until PCR positive for presence of malaria parasites). Once PCR positive they will be monitored twice-daily morning (AM) and evening (PM) until treatment, for adverse events and the unexpected early onset of symptoms, signs or parasitological evidence of malaria. On the day designated for commencement of treatment as determined by qPCR results (approximately Study day 7), participants will be admitted to the study unit and monitored. The threshold for commencement of treatment will be when PCR quantification of all participants is = 5,000 parasites/mL. If the PCR quantification of any participant is = 5,000 parasites/mL and is accompanied by a clinical symptom score >5, before all participants have reached the treatment threshold (PCR quantification of = 1,000), then treatment of that participant will begin within a 24 h period. Participants will be followed up as inpatients for at least 48 h to ensure tolerance of the treatment and clinical response, then if clinically well on an outpatient basis for safety and clearance of malaria parasites via PCR.

Cohort1. Following initial piperaquine treatment, a repeat dose of piperaquine (960 mg) may be administered on an outpatient basis if recrudescent asexual parasitemia occurs (defined as 3 consecutively increasing parasite count over 1000 parasites/mL). Participants will also be evaluated for the presence of gametocytes in the blood, as determined by qPCR (amplification of pfs25 gametocyte-specific transcript). Assessment of OZ439 gametocytocidal properties and transmission studies will be undertaken when gametocytemia appears. Participants will be randomised into an experimental or a control group when peak gametocytemia occurs (approximately 15 days after administration of piperaquine i.e. about day 22 of the study). Participants in the experimental group (n=2 per dose cohort) will be administered OZ439 as a single 500 mg dose and participants in the control group (n=2) will receive primaquine 15 mg as a single dose. Blood will be collected (AM) from each participant in both groups for membrane feeding assays with An. stephensi vector mosquitoes. For direct feeding assays (DFA), participants will be escorted to the quarantine insectary facility at QIMR Berghofer Medical Research Institute and asked to allow vector mosquitoes to feed on the volar surface of their forearms, calves or thighs for a period of 10 ± 5 minutes. The experimental infection of mosquitoes by direct feeding on participants will be performed up to a maximum of three time points over a maximum interval of up to 10 days, approximately 15 days post-piperaquine treatment (1 direct feed prior to receiving OZ439 (active) or primaquine (control), and 2 feeds scheduled following OZ439 (active) or primaquine (control) treatment). Artificial (indirect) membrane feeding (IFA) may occur up to 10 times prior to curative anti-malarial treatment at the End of Study with Riamet® (artemether-lumefantrine)and primaquine (45 mg).

Cohort2 and 3. A similar study design and treatment procedure will be used for the two subsequent cohorts. Doses of OZ439 to be evaluated will be selected after analysis of the data from cohort1. Doses of OZ439 will not exceed 1200 mg.

Pre-emptive rescue treatment with Riamet® can commence whenever deemed necessary by the investigator. Participants can be administered the rescue Riamet® on site for initial dosing followed by monitoring, either in clinic, or by telephone for three days to ensure adherence to Riamet® therapy.

Participants will be treated with a single dose of primaquine (45 mg) as described in section 4.4.2 in this protocol concurrent with their Riamet® treatment to ensure clearance of any gametocytes present.

Adverse events will be monitored via telephone monitoring, within the clinical research unit, and on outpatient review after malaria challenge inoculation and anti-malarial study drugs administration. Blood samples for safety evaluation, malaria monitoring, and red blood cell antibodies will be drawn at screening.

ELIGIBILITY:
Inclusion Criteria:

Demography:

* Adult (male and females) participants between 18 and 55 years of age, inclusive who do not live alone (from Day 0 until at least the end of the anti-malarial drug treatment) and be contactable and available for the duration of the trial (maximum of 6 weeks).
* Body weight, minimum 50.0 kg, body mass index between 18.0 and 32.0 kg/m

Health status:

* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 10 minutes resting in supine position:
* 90mmHg < systolic blood pressure (SBP) <140 mmHg,
* 50 mmHg < diastolic blood pressure (DBP) <90 mmHg,
* 40 bpm< heart rate (HR) <100 bpm.
* Normal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position, QTcF=450 ms average with absence of second or third degree atrioventricular block or abnormal T wave morphology.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy participants enrolled in this clinical investigation. More specifically for serum creatinine, hepatic transaminase enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the Participant has documented Gilbert syndrome) should not exceed the upper laboratory norm and haemoglobin must be equal or higher than the lower limit of the normal range, - - As there is the risk of adverse effects of OZ439, Riamet and primaquine in early pregnancy, it is important that any participants involved in this study do not get pregnant or get their female partners pregnant.

Regulations:

- Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

Medical history and clinical status:

* Any history of malaria or participation to a previous malaria challenge study
* Must not have travelled to or lived (>2 weeks) in a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.
* Known severe reaction to mosquito bites other than local itching and redness
* Has evidence of increased cardiovascular disease risk (defined as >10%, 5 year risk) as determined by the method of Gaziano et al. (1). Risk factors include sex, age, systolic blood pressure (mm/Hg), smoking status, body mass index (BMI, kg/m) and reported diabetes status.
* History of splenectomy.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician or history of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion.
* Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunodeficiencies), insulin-dependent and NIDDM diabetes (excluding glucose intolerance if E04 is met ), progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, psoriasis, rheumatoid arthritis, asthma, epilepsy or obsessive compulsive disorder, skin carcinoma excluding non-spreadable skin cancers such as basal cell and squamous cell carcinoma
* Participants with history of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis including depression or receiving psychiatric drugs or who has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Frequent headaches and/or migraine, recurrent nausea, and/or vomiting (more than twice a month).
* Presence of acute infectious disease or fever (e.g., sub-lingual temperature = 38.5°C) within the five days prior to inoculation with malaria parasites.
* Evidence of acute illness within the four weeks before trial prior to screening that the Investigator deems may compromise subject safety.
* Significant intercurrent disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.
* Participant has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion, e.g. gastrectomy, diarrhoea.
* Participation in any investigational product study within the 12 weeks preceding the study.
* Blood donation, any volume, within 1 month before inclusion or participation in any research study involving blood sampling (more than 450 mL/ unit of blood), or blood donation to Red Cross (or other) blood bank during the 8 weeks preceding the reference drug dose in the study.
* Participant unwilling to defer blood donations for 6 months.
* Medical requirement for intravenous immunoglobulin or blood transfusions.
* Participant who has ever received a blood transfusion.
* Symptomatic postural hypotension at screening, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure =20 mmHg within 2-3 minutes when changing from supine to standing position.
* History or presence of alcohol abuse (alcohol consumption more than 40 g per day) or drug habituation, or any prior intravenous usage of an illicit substance.
* Smoking more than 5 cigarettes or equivalent per day and unable to stop smoking for the duration of the study.
* Ingestion of any poppy seeds within the 24 hours prior to the screening blood test (participants will be advised by phone not to consume any poppy seeds in this time period).

Interfering substance:

* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life (whichever is longer) of the medication,
* Any vaccination within the last 28 days.
* Any corticosteroids, anti-inflammatory drugs, immunomodulators or anticoagulants. Any participant currently receiving or having previously received immunosuppressive therapy, including systemic steroids including adrenocorticotrophic hormone (ACTH) or inhaled steroids in dosages which are associated with hypothalamic-pituitary-adrenal axis suppression such as 1 mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids (budesonide 800 µg per day or fluticasone 750 µg).
* Any recent or current systemic therapy with an antibiotic or drug with potential anti-malarial activity (chloroquine, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, hydroxychloroquine, etc.).

General conditions:

* Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any participant in the exclusion period of a previous study according to applicable regulations.
* Any participant who lives alone (from Day 0 until at least the end of the anti-malarial drug treatment).
* Any participant who cannot be contacted in case of emergency for the duration of the trial and up to 2 weeks following end of study visit.
* Any participant who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
* Any participant without a good peripheral venous access.

Biological status:

* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, antihepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab),
* Participant is found to be G6PD deficient.
* Any drug listed in Table 2 in the urine drug screen unless there is an explanation acceptable to the medical investigator (e.g., the participant has stated in advance that they consumed a prescription or OTC product which contained the detected drug) and/or the Participant has a negative urine drug screen on retest by the pathology laboratory.
* Positive alcohol - breath test.

Specific to the study:

* Cardiac/QT risk:

  * Known pre-existing prolongation of the QTc interval considered clinically significant
  * Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc-interval or any clinical condition known to prolong the QTc interval. History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
* Known hypersensitivity to OZ439, piperaquine or any of its excipients or 4-aminoquinolines, artemether or other artemisinin derivatives, lumefantrine, or other arylaminoalcohols.
* Unwillingness to abstain from quinine containing foods/beverages such as tonic water, lemon bitter, from inoculation (Day 0) to the end of the malaria treatment.
* Any history or presence of lactose intolerance.

On dosing day, and during the blood collection intervals:

* Ingestion of any other drug, in the two weeks prior to dosing or during the blood sampling period that, in the opinion of the Medical Investigator, could compromise the study, e.g., through pharmacokinetic or metabolic interactions, or analytical interference. However the Medical Investigator may permit the use of paracetamol for the treatment of headache or other pain. If drug therapy other than paracetamol or drug specified in the protocol, is required during the study periods, a decision to continue or discontinue the participant's participation will be made by the Medical Investigator, based on the nature of the medication and the time the medication was taken.
* Failure to conform to the requirements of the protocol.
* Detection of any drug listed in this protocol in the urine drug screen unless there is an explanation acceptable to the medical investigator (e.g., the participant has stated in advance that they consumed a prescription or OTC product which contained the detected drug).
* Vital signs outside the reference range and considered as clinically significant by the Investigator or his representative.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, Prof, Principal Investigator — QIMR Berghofer Medical Research Institute
Locations (1):
- Q-Pharm Clinics, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collins KA, Wang CY, Adams M, Mitchell H, Rampton M, Elliott S, Reuling IJ, Bousema T, Sauerwein R, Chalon S, Mohrle JJ, McCarthy JS. A controlled human malaria infection model enabling evaluation of transmission-blocking interventions. J Clin Invest. 2018 Apr 2;128(4):1551-1562. doi: 10.1172/JCI98012. Epub 2018 Mar 12. PMID 29389671

RESULTS

PARTICIPANT FLOW:
Groups:
- Primaquine 15mg: Administration of Primaquine 15mg (control).
  Each participant in the cohort will be inoculated on Day 0 with ~2,800 viable parasites of Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. When PCR quantification of all participants is ≥ 5,000 parasites/mL, they will receive a single dose of 480 mg of piperaquine phosphate to clear blood stage parasitemia. When gametocytemia is at the peak (approximately 15 days after administration of piperaquine), participants of this arm will receive 15mg of Primaquine treatment as the control.
- OZ439 500mg: Administration of OZ439 500mg.
  Each participant in the cohort will be inoculated on Day 0 with ~2,800 viable parasites of Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. When PCR quantification of all participants is ≥ 5,000 parasites/mL, they will receive a single dose of 480 mg of piperaquine phosphate to clear blood stage parasitemia. When gametocytemia is at the peak (approximately 15 days after administration of piperaquine), participants will receive 500mg of OZ439.
Period: Overall Study
Arm/Group | Primaquine 15mg | OZ439 500mg
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primaquine 15mg | OZ439 500mg | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (5.1) | 29.2 (12.97) | 28.2 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (3.68) | 23.68 (2.902) | 24.96 (3.434)

OUTCOME MEASURES:

1. Primary Outcome: Infection Success of Vector Mosquitoes
Description: Assessing the transmissibility by oocyst detection in mosquito midgut preparations following direct and membrane (indirect) feeding.
Time Frame: From day 10 to 21 post Piperaquine dosing
Population: Transmission of gametocytes to mosquitos was only determined for 7 of the 11 subjects that participated in the trial. Transmission of gametocytes to mosquitoes was observed in 5 of the 7 subjects analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Primaquine 15mg | OZ439 500mg
Number analyzed (Participants) | 3 | 4
Participants | 2 | 3

2. Secondary Outcome: Safety: Number of AEs
Description: Adverse events incidence
Time Frame: From Challenge inoculum on day 0 until end of study on day 31
Measure: Number; unit: Number of adverse events
Arm/Group | Primaquine 15mg | OZ439 500mg
Number analyzed (Participants) | 5 | 6
Number of adverse events | 17 | 4

ADVERSE EVENTS:
Time Frame: Until end of study on Day 34 (Cohort 1) or Day 36 (End of Study visit for cohorts 2a, 2b, and 3).
Arm/Group | Primaquine 15mg | OZ439 500mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 4/5 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primaquine 15mg (N=5) | OZ439 500mg (N=6)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyperhidrosis (General disorders) | 1 (1) | 0 (0)
Lethargy (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Puncture site reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less